CLINICAL TRIAL: NCT03038919
Title: Pilot Randomized, Controlled Trial of Testosterone Therapy in Chronic Critically Ill Patients and Its Potential Effects on Weaning From Mechanical Ventilation and Intensive Care Unit-acquired Weakness
Brief Title: Role of Anabolic Steroids on Intensive Care Unit-Acquired Weakness
Acronym: RAS-ICU
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0293
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Critical Illness Polyneuropathies
Keywords: prolonged mechanical ventilation; critically ill patients; anabolic steroid
MeSH Terms: conditions — Polyneuropathies | interventions — testosterone 17 beta-cypionate; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anabolic patients (Experimental): Intramuscular injection of testosterone cypionate 200mg every 15 days in addition to standard nutrition and physical therapy at ICU.
  Interventions: Drug: Testosterone cypionate; Other: Standard nutrition and physical therapy at ICU
- Control (Other): Standard nutrition and physical therapy at ICU without administration of testosterone cypionate
  Interventions: Other: Standard nutrition and physical therapy at ICU

INTERVENTIONS:
Drug: Testosterone cypionate — Bi-weekly intramuscular injection of testosterone cypionate 200mg.
  Other Names: testosterone
  Arms: Anabolic patients
Other: Standard nutrition and physical therapy at ICU — follow-up of the patient without use of testosterone cypionate

SUMMARY:
The researchers intend to investigate possible anabolic effects of bi-weekly exogenous testosterone administration during intensive care unit (ICU) stay for up to 8 weeks. Control group will receive standard ICU management and will also be followed during ICU stay.

DETAILED DESCRIPTION:
For the study chronic critical patients will be included according to criterion of mechanical ventilation by orotracheal tube> 14 consecutive days or mechanical ventilation by tracheostomy> 8 consecutive days and that do not present exclusion criteria.

Patients will be randomized into two follow-up groups: Intervention group with anabolic steroid and control group.

The anabolic steroid intervention group will receive a bi-weekly dose of 200mg intramuscular testosterone cypionate and receive the standard treatment of nutritional therapy and physical therapy. While patients in the control group will receive only the standard treatment of nutrition and physical therapy, without addition of the anabolic drug.

At the beginning of the study and weekly the patients will be evaluated in relation to the muscular profile with diaphragm ultrasound and Medical Research Council (MRC) application. In addition to the collection of serum homograms, leukogram, lipid profile and renal function tests.

Weight and nutritional therapy-related data will be identified in the patient's chart regarding caloric and protein requirement and supply adequacy.

In the inclusion and biweekly will be collected serum levels of free testosterone, blood count, leukogram, blood gas, renal function and liver function. Nitrogen balance of patients from urinary urea will be performed.

The evaluations of the groups and the intervention with the anabolic steroid will be of 8 weeks or during the period of dependence of the mechanical ventilation. After this period the patients will be monitored for the outcome: length of stay in the intensive care unit, hospital stay until discharge and clinical outcome: death or discharge.

ELIGIBILITY:
Inclusion Criteria:

* Individuals older than 18 years
* Mechanical ventilation by orotracheal tube for more than 14 consecutive days
* Mechanical ventilation by tracheostomy for more than 8 consecutive days

Exclusion Criteria:

* End of life care
* Known hypersensitivity to formula
* Venous or arterial thrombosis within last 6 months: ischemic stroke, myocardial infarction, acute peripheral arterial occlusion, acute mesenteric ischemia, deep venous thromboembolism, pulmonary embolism
* Decompensated congestive heart failure
* Acute liver failure or acute on chronic liver failure
* Refractory shock (norepinephrine dose >0.3 mcg/kg/min or equivalent doses of any vasoactive agent)
* Platelets below <20,000 / mm3 without transfusion plan
* Personal history of prostate cancer
* Primary neuromuscular disorders such as myasthenia gravis, Guillain-Barré syndrome, amyotrophic lateral sclerosis, Duchenne Muscular dystrophy
* Current or prior spinal cord injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation dependence | 8 weeks
  Days of any positive pressure ventilation described in the patient record from the start of the study

SECONDARY OUTCOMES:
Muscle weakness | 8 weeks
  The muscle weakness measured weekly by the study team through the Medical Research Council (MRC)
Ultrasound diaphragm | 8 weeks
  Weekly the study team will perform diaphragm ultrasound to monitor the respiratory muscles, observing measures of inspiration and expiration.
ICU length of stay | 9 months
  Patient's length of stay in the intensive care unit after the start of the study as described in the patient record
Hospital length of stay | 9 months
  Period of stay of the patient in the hospital after discharge from the intensive care unit described in the patient record

CONTACTS AND LOCATIONS:
Overall Officials: Silvia RR Vieira, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre - RS
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided